CLINICAL TRIAL: NCT05262686
Title: Efficacy and Immunological Evaluation of Belimumab Plus Low Dose IL-2 in the Treatment of Systemic Lupus Erythematosus: a Randomised Prospective Study
Brief Title: Efficacy and Immunological Evaluation of Belimumab Plus Low Dose IL-2 in the Treatment of Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Peking2021SLE
Record Dates: First submitted 2022-02-22; First posted 2022-03-02 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- belimumab plus low dose IL-2 (Experimental): 10mg/kg belimumab was intravenously injected to patients with systemic lupus erythematosus every month for 24 weeks.
  Interleukine-2 was first added to the original treatment for systemic lupus erythematosus with 1 million IU qod for 12 weeks, injected subcutaneously at the outer side of upper arm, abdomen and thigh, then the same dose of IL-2 was injected once a week for 12 weeks subcutaneously.
  Interventions: Drug: Belimumab; Drug: Interleukin-2
- belimumab (Active Comparator): 10mg/kg belimumab was administrated to patients with systemic lupus erythematosus for at least 24 weeks, intravenously injected every month.
  Interventions: Drug: Belimumab
- low dose IL-2 (Active Comparator): The first stage: interleukine-2 was added to the original treatment for systemic lupus erythematosus with 1 million IU qod for 12 weeks, injected subcutaneously at the outer side of upper arm, abdomen and thigh; The second stage: 1 million IU IL-2 was injected once a week for 12 weeks subcutaneously.
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Belimumab — Belimumab was intravenously administrated at a dose of 10mg/kg once a month for at least 24 weeks.
  Arms: belimumab; belimumab plus low dose IL-2
Drug: Interleukin-2 — Low lose interleukine-2 at a dose of 1 million IU was injected once every other day for 12 weeks, then the same dose of IL2 was injected once a week at the second stage for 12 weeks.
  Other Names: Recombinant Human interleukine-2
  Arms: belimumab plus low dose IL-2; low dose IL-2

SUMMARY:
The purpose of this study was to explore the clinical and immunological efficacy of belimumab plus low dose IL-2 in systemic lupus erythematosus.

DETAILED DESCRIPTION:
Given that belimumab and low dose interleukin-2 (IL-2) have been widespreadly applied in the treatment of systemic lupus erythematosus (SLE), this study designed a randomised, single center, prospective study to investigate the effects and safety of combined utilization of belimumab and low dose IL-2. SLE patients were allocated in each group randomly (n=10) and regularly administered belimumab (10mg/kg) with or without IL-2 (1 million IU). Then, we evaluated the improvement of clinical and laboratory indexes and monitored the changes of immune cell subsets and cytokines.

ELIGIBILITY:
Inclusion Criteria:

- 1. Male or female >18 years of age at screening visits 2. Patients meet the American-European Consensus Group 2002 classification criteria 3. The patient must be informed in writing of the consent to participate in the trial and the patient is expected to be able to comply with the requirements of the study follow-up plan and other protocols.

4. Dosing of antimalarials, prednisone or equivalent, cholinergic stimulants, and topical cyclosporine required to be stable for at least 4 weeks before screening and during study; maximum doses allowed:

* Hydroxychloroquine, 400 mg/day;
* Prednisone, 10 mg/day

Exclusion Criteria:

* 1. Any subject meeting any of the following criteria should be excluded: 1. Laboratory abnormality: • Hb≤9 g/dl • Neutrophil 10 mg/d) within 1 month.

  2. Serious complications: including heart failure (≥ New York Heart Association (NYHA) class III), renal insufficiency (creatinine clearance ≤ 30 ml/min), liver dysfunction (serum Alanine transaminase (ALT) or aspartate aminotransferase (AST) greater than three times the upper limit of normal, or total bilirubin greater than Normal upper limit) 3. Known allergies, hyperreactivity or intolerance of tofacitinib or its excipients.

  4. Have a serious infection needing hospitalization (including but not limited to hepatitis, pneumonia, bacteremia, pyelonephritis, Epstein-Barr virus (EBV), tuberculosis infection), or use intravenous antibiotics to treat infection in 2 months before the enrollment.

  5. Infection with HIV (HIV antibody positive serology) or hepatitis C (Hep C antibody positive serology). If seropositive, it is recommended to consult a doctor who has expertise in treating HIV or hepatitis C virus infection.

  6. Any known history of malignancy in the past 5 years (except for nonmelanoma skin cancer, non-melanoma skin cancer or cervical tumor without recurrence within 3 months after surgical cure prior to the first study preparation).

  7. Uncontrolled mental or emotional disorders, including a history of drug and alcohol abuse over the past 3 years, may hinder the successful completion of the study.

  8. Pregnant, lactating women (WCBP) are reluctant to use medically approved contraceptives during treatment and 12 months after treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Immunological responses of B cell subsets | Week 24
  A significant reduction of active B cell subsets including naive B cells and transitional B cells after different interventions. P values below 0.05 are considered statistically significant in this study.

SECONDARY OUTCOMES:
Proportion of SLE Responder Index (SRI)4 response | Week 12 and 24
  SLE Responder Index (SRI)4 responders had ≥4-point reduction in safety of estrogens in Lupus Erythematosus National Assessment-SLE Disease Activity Index(SELENA-SLEDAI) score
Prednisone dose | Week 12 and 24
  The improvement in prednisone dose experienced a mean corticosteroid dose reduction of ≥25% mg/day at baseline to ≤7.5 mg/day.
Immunoglobulin change from baseline | Week 12 and 24
  Serum samples were collected at indicated time-points for analysis of immunoglobulins: Immunoglobulin G (IgG), Immunoglobulin A (IgA), and Immunoglobulin M (IgM). Baseline is defined as the Day 0 visit from parent studies.
Autoantibody change from baseline | Week 12 and 24
  Blood samples were collected at indicated time-points for analysis of autoantibodies like anti-double stranded deoxyribonucleic Acid(dsDNA), antinuclear antibody (ANA). Baseline is defined as the Day 0 visit from parent studies.
Change of complement C3 and C4 Levels from baseline | Week 12 and 24
  Blood samples were collected at indicated time-points for analysis of complement levels like complement 3 (C3) and complement 4 (C4). Baseline is defined as the Day 0 visit from parent studies.
Safety and tolerability of the treatment | Up to Week 24
  The incidence of adverse events, disease activity and clinical laboratory data throughout the study were accessed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Peking University Institute of Rheuamotology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, China